CLINICAL TRIAL: NCT05687110
Title: A Phase 1 Study of the Polymerase Theta (POLθ) Inhibitor Novobiocin in BRCA- Mutant and Other DNA Damage Repair-Deficient Solid Tumors
Brief Title: Studying the Safety and Determining the Optimal Dose of Novobiocin in Patients With Tumors That Have Alterations in DNA Repair Genes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-06608; NCI-2022-06608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DF/HCC 23-235; 10528 (Other: Dana-Farber - Harvard Cancer Center LAO); 10528 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2023-01-14; First posted 2023-01-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; X-Rays; Novobiocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (novobiocin sodium) (Experimental): Patients receive novobiocin sodium PO QD for 5 days in a row followed by 2 days off each week. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy, medical imaging scans, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging Testing; Biological: Novobiocin Sodium

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Diagnostic Imaging Testing — Undergo medical imaging scans
  Other Names: Diagnostic Imaging; Medical Imaging
Biological: Novobiocin Sodium — Given PO

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of novobiocin in treating cancer patients with alterations in deoxyribonucleic acid (DNA) repair genes. Novobiocin is an antibiotic that blocks the activity of a protein called DNA polymerase theta, which helps repair DNA that has become damaged as cells grow and divide. Cancer cells that cannot repair their damaged DNA die. This medication may help shrink or stabilize cancer with a mutation in DNA repair genes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of novobiocin sodium (novobiocin) administered on a 5-days on/2-days off schedule in patients with solid tumors carrying homologous recombination (HR) or DNA damage repair (DDR) alterations that are poly (ADP-ribose) polymerase (PARP) inhibitor-naïve or -resistant.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the safety and tolerability of novobiocin administered on a 5-days on/2-days off schedule in patients with solid tumors carrying HR or DDR alterations that are PARP inhibitor-naïve or -resistant.

III. To characterize the pharmacokinetic parameters of novobiocin administered on a 5-days on/2-days off schedule in patients with solid tumors carrying HR or DDR alterations that are PARP inhibitor- naïve or -resistant.

IV. To determine the minimally biologically effective dose of novobiocin in patients with solid tumors carrying HR or DDR alterations that are PARP inhibitor-naive or -resistant using pre- and on-treatment biopsies to characterize novobiocin-mediated pharmacodynamic effects.

V. To conduct a preliminary assessment of anti-tumor activity of novobiocin administered on a 5-days on/2-days off schedule.

EXPLORATORY OBJECTIVES:

I. Whole exome sequencing (WES) of pre- and time-of-progression biopsies to characterize tumors for HR deficiency (deleterious mutations/deletions in genes known to be involved in HR) and genomic changes mediating acquired resistance to novobiocin.

II. Ribonucleic acid sequencing (RNAseq) on pre- and on-treatment biopsies, as well as time-of-progression biopsies for serial analysis of gene expression to identify determinants of response, resistance, and pathway adaptation to novobiocin.

III. Correlation of baseline level of POLQ messenger ribonucleic acid (mRNA) with clinical outcome (complete response [CR], partial response [PR] or stable disease [SD] versus [vs.] progressive disease [PD]).

IV. Correlation of ATM immunohistochemistry (IHC) with clinical outcome in patients with ATM-mutant cancers.

OUTLINE: This is a dose-escalation study.

Patients receive novobiocin sodium orally (PO) once daily (QD) for 5 days in a row followed by 2 days off each week. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy, medical imaging scans, and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have histologically confirmed solid tumor with a known pathogenic mutation in BRCA1/2, PALB2, RAD51C, RAD51D, ATM, BARD1, BLM, BRIP1, CDK12, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, NBN (NBS1), RAD50 and RAD51B as confirmed by a Clinical Laboratory Improvement Amendments (CLIA)-certified method. Patients with alterations defined only by germline testing are eligible. Other qualifying HRD alterations may be considered if approved by the principal investigator and the Cancer Therapy Evaluation Program (CTEP) monitor
* Any number of prior therapy regimens is allowed
* Patients with cancers for which PARP inhibitors have been approved as standard-of-care must have received a PARP inhibitor prior to enrollment on this study. Other patients may be either PARP inhibitor-naïve (i.e., never have received a PARP inhibitor) or have disease that is PARP inhibitor-resistant (i.e., disease that has progressed radiologically based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 while receiving any PARP inhibitor)
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of novobiocin in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group Performance (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Leukocytes >= 3,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN)
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine transferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 1.5 × institutional ULN
* Glomerular filtration rate (GFR) >= 60 mL/min (via the chronic kidney disease epidemiology [CKD-EPI] glomerular filtration rate estimation)
* Fridericia's formula-corrected QT interval (QTcF) =< 480 ms
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression, stable and off steroids for 1 month
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the patient is asymptomatic and the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients should be New York Heart Association Functional Classification of class 2B or better
* Patients must have tumors amenable to biopsies, and be willing to undergo biopsies at two time points (pre- and on-treatment)
* The effects of novobiocin on the developing human fetus are unknown. For this reason and because polymerase theta (POLtheta) inhibitor agents have the potential to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 4 months after completion of novobiocin administration. Effective contraception is defined as a method that achieves a failure rate of less than 1% per year when used consistently and correctly. (Note: Because of a concern for decreased effectiveness of estrogen-containing oral agents when given with novobiocin, barrier methods and abstinence are the preferred methods for contraception). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to novobiocin
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4/5 are ineligible. Patients receiving any medications or substances that are known to be substrates of breast cancer resistance protein (BCRP/ABCG2) and/or organic anion transporting polypeptides (OATP1B1, OATP1B3 and OATP2B1) and/or organic anion transporters (OAT1 and OAT3) within 14 days prior to the first dose of study drug are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients using herbal/dietary supplements with known hepatotoxicity risk are ineligible
* Patients receiving concurrent medications associated with a risk of corrected QT interval (QTc) prolongation and/or Torsades de Pointes are not allowed within 14 days of initiation of study treatment. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference such as CredibleMeds or Lexicomp. Drugs listed in the "drugs to avoid in CLQTS (congenital long QT syndrome)" and "known risk of TdP (torsade de pointes)" should be excluded. Granisetron is an acceptable antiemetic on this study. If a patient must take ondansetron, they may NOT take any other concomitant agents which might impact their QTc
* Patients must have UGT1A1 testing at screening. Patients homozygous for A(TA)7TAA in the promoter region (also known as UGT1A1 *28), homozygous for the G71R allele (also known as UGT1A1*6), or with compound alterations of *28 and *6, are excluded as they are at risk for further reduction of UGT1A1 activity that may disrupt bilirubin clearance

  * UGT1A1 testing must address both *28 and *6 alterations
* Patients with uncontrolled intercurrent illness. Additionally, patients with acute liver disease, poorly controlled liver disease, or cirrhosis are excluded
* Patients with (known) active or poorly controlled alcohol use disorder are excluded
* Pregnant women are excluded from this study because novobiocin is a POLtheta inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with novobiocin, breastfeeding should be discontinued if the mother is treated with novobiocin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase 2 dose of continuous novobiocin administration | Up to 2 years
  The MTD will be identified as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. Standard hematological and non-hematologic parameters, scored using Common Terminology Criteria for Adverse Events version 5.0, will be used to define dose limiting toxicity.

SECONDARY OUTCOMES:
Radiological response | Up to 2 years
  Radiological response will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1 criteria and will be graded as complete response (CR), partial response (PR), stable disease (SD) and progressive disease.
Response rate | Up to 2 years
  Response rate (CR + PR) will be summarized by frequencies and percentages, by dose level.
Clinical benefit rate | Up to 2 years
  Clinical benefit rate (CR + PR + SD > 24 weeks) will be summarized by frequencies and percentages, by dose level.
Progression free survival | From study enrollment until the identification of disease progression or death, assessed up to 2 years
  Will be summarized using Kaplan-Meier curves by dose-level (for dose levels with sufficient sample size to permit estimation).
Median duration of response | Up to 2 years
  Median duration of response will be reported with ranges.
Plasma concentrations of novobiocin | Days 1 & 17 of cycle 1 (pre-treatment and 0.5, 1, 2, 4, 6, 8, & 24 hours post-treatment) and days 2 & 25 of cycle 2 (pre-dose and 24 hours post-treatment)
  Will be quantitatively measured using liquid chromatography with tandem mass spectrometry to derive standard pharmacokinetic parameters.
Biological effectiveness | Up to 2 years
  Biological effectiveness will be defined as an increase in the percentage of RAD51-foci positive cells (> 5 foci/nucleus) from =< 10% on the pre-treatment biopsy to >= 30% at the on-treatment biopsy in patients with poly (ADP-ribose) polymerase inhibitor-resistant tumors. A biologically effective dose will be one that induces an increase in gamma-H2AX in the on-treatment compared to the pre-treatment biopsy.

OTHER OUTCOMES:
POLQ messenger ribonucleic acid level (mRNA) | Up to 2 years
  Other pharmacodynamic data will be captured using descriptive statistics. In an exploratory fashion, will analyze correlations between baseline POLQ mRNA level and clinical outcome.
ATM immunohistochemistry (IHC) | Up to 2 years
  Other pharmacodynamic data will be captured using descriptive statistics. In an exploratory fashion, will analyze correlations between ATM IHC and genomic alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey I Shapiro, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (23):
- United States (22):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm